CLINICAL TRIAL: NCT02918903
Title: Evaluation of Pulpal Symptoms Following Minimal Caries Removal Technique in Comparison to Complete Caries Removal in Molars With Deep Caries
Brief Title: Evaluation of Pulp Symptoms After Minimal Caries Removal in Treatment of Deep Caries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nouran Mamdouh Ahmed, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEBD-CU-2016-09-206
Record Dates: First submitted 2016-09-26; First posted 2016-09-29 (Estimated); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Deep Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Minimal caries removal (Experimental): the patients in this group will be treated by minimal caries removal technique, where only caries at lateral walls of cavity is removed, stainless steel crown preparation is performed and then stainless steel crown is placed as final restoration.
  Interventions: Procedure: Minimal caries removal
- Complete caries removal (Active Comparator): patients in this group will be treated by complete caries removal technique, where all caries will be removed, a base of resin modified glass ionomer is placed and then stainless steel crown is placed as final restoration.
  Interventions: Procedure: Complete caries removal

INTERVENTIONS:
Procedure: Minimal caries removal — the experimental group will be treated by minimal caries removal where only caries at lateral walls of cavity will be removed then stainless steel crown will be placed as final restoration.
  Arms: Minimal caries removal
Procedure: Complete caries removal — the control group will be treated by complete caries removal where all caries along lateral and pulpal walls of cavity will be removed, a base of resin modified glass ionomer will be placed then stainless steel crown will be placed as final restoration.
  Arms: Complete caries removal

SUMMARY:
The objective of this study is to assess and compare the possible post-operative pulpal symptoms (Spontaneous pain, pain on percussion, swelling, sinus or fistula), incidence of pulp exposure, child acceptance, chair time and radiographic success between two techniques for managing dental caries: minimal caries removal and complete caries removal in primary molars.

DETAILED DESCRIPTION:
Minimal Caries Removal (MCR) technique was described in 2015 by Chompu-inwai et al., as a treatment option for primary molars with deep carious lesions or reversible pulpitis where only soft demineralized dentin around the lateral walls of the carious lesion is removed. The aim of this study is to assess the success of such a technique in managing primary molars with asymptomatic deep caries in terms of; post-operative pulpal symptoms(spontaneous pain, pain on percussion, fistula or sinus), incidence of pulp exposure, child acceptance, chair time and radiographic success.

ELIGIBILITY:
Inclusion Criteria:

* Primary molar with deep dentin caries involving occlusal &/or occluso-proximal surfaces.
* Absence of clinical signs and symptoms of irreversible pulpitis such as spontaneous pain. Only presence of pain provoked with stimulation, such as complaints of food impaction when eating is allowed.
* Absence of clinical swelling or pus exudates/fistula of soft or periodontal tissues.
* Absence of abnormal tooth mobility.
* Absence of pain on percussion.
* Restorable tooth.

Radiographic inclusion criteria:

* Extension of dental caries one-third or more of the entire dentin thickness.
* No super- imposition of dental caries on the dental pulp.
* No widened periodontal ligament (PDL) space.
* No radiolucency in the peri-apical or furcation areas.
* No pathologic internal or external root resorption.
* No pulp canal calcification or obliteration.

Exclusion Criteria:

1. Patients experience any signs or symptoms of pulpal or peri-apical pathology.
2. Patients with systemic diseases requiring special dental consideration.
3. Unmotivated, uncooperative patients.
4. Patients unable to attend follow-up visits.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Post operative pain assessed by direct questioning as binary outcome | 9 months
  Assessed by direct questioning pain history

SECONDARY OUTCOMES:
incidence of pulp exposure | Within 30 minutes
  The outcome will be measured during the treatment visit which is estimated to be 30 minutes
radio-graphic success | 9 months
  No external or internal root resorption, no periapical or furcation radiolucencies, no widening of periodontal membrane space

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of denntistry, Cairo, El-manyal, Egypt

IPD SHARING:
Plan to Share IPD: No